CLINICAL TRIAL: NCT02268487
Title: THE AIUNI - Integral Assessment in Unipolar Depression
Brief Title: Integral Assessment in Unipolar Depression
Acronym: AIUNI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., Fernando Fernandes, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 795996
Record Dates: First submitted 2014-10-08; First posted 2014-10-20 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Major Depressive Disorder
Keywords: Early Improvement; Depression; Antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sertraline (Experimental): Patients using Sertraline with any dose will be evaluated about Early Improvement
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Treatment
  Other Names: Early Improvement

SUMMARY:
The objective of this project is to assess the occurrence of early improvement within the first two weeks of antidepressant treatment and to correlate this improvement with favorable therapeutic outcome at the end of the acute and treatment continuation phases (8 and 24 weeks, respectively).

DETAILED DESCRIPTION:
An ongoing debate, as long-running as treatment with antidepressants itself, is the delay in response to these drugs. Antidepressant drugs take 2 to 4 weeks to produce the treatment response effect (at least 50% improvement in depressive symptoms versus baseline levels). This delay in antidepressant response can prove highly problematic since, during this interim period, the patient is exposed to the suffering, debilitative effects, direct and indirect costs and risks associated with major depressive disorder (MDD).

Another important issue is when to define failure of a therapeutic trial and how to change treatment. Between 30 and 50% of MDD patients fail to respond to adequate first-line treatment. If favorable outcome is defined as full remission (as opposed to only 50% improvement) of the patient, the failure rate during first trial is greater still. Some reviews recommend dose adjustments every two weeks and a 4-8 week wait before treatment change for poor response. Despite these recommendations, the question over when and how to change treatment strategy warrants further debate.

Early improvement in antidepressant treatment is desirable because it reduces the suffering, losses and costs associated with MDD. In addition, the risk of suicidal ideation or committing suicide are reduced in patients presenting early improvement of depressive symptoms. However, early improvement not only reduces risk but also predicts outcome at the end of the acute phase of treatment. A number of studies investigating different antidepressants have shown that the presence of early response is a good predictor of favorable outcome at the end of the acute phase of treatment (after 6 or 8 weeks of treatment). A meta-analysis reviewing 41 simple or double-blind clinical trials included a total of 6562 patients.

Early improvement, defined as a 20% reduction in score on the Hamilton Depression Scale (HAMD-17) within 2 weeks, was associated with sustained response, remission (defined as HAM-D-17 score ≤7). While early response has been amply demonstrated in numerous clinical trials, there are gaps in knowledge on the subject. Scant studies have documented whether there are differences in the pattern of early improvement among different antidepressants. Similarly, there is a dearth of studies analyzing whether the presence or otherwise of early response has the same predictive value for different antidepressants. Another little explored aspect is the arbitrary nature of the criteria defining onset of improvement, early improvement, treatment response and symptomatological remission. Studies tend to reproduce previously-adopted criteria without elaborating on the exploratory analyses justifying the cut-off points adopted.

The aim of the present study is to assess the presence of early improvement after one and two weeks of treatment with sertraline. Besides assessing the presence of early response, the study will include an exploratory analysis assessing positive and negative predictive values, sensitivity and specificity of early improvement as a predictor of sustained response and remission after 6, 8 and 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients Presenting Depressive Episode according to DSM-IV-TR

Exclusion Criteria:

* Patients presenting: psychotic symptoms, Axis 1 comorbidities (except specific phobia, specific social phobia and nicotine dependence) or risk of suicide (defined as score = 3 on item 3 of the 17-item HAMD or at the discretion of rater);
* Other exclusion criteria are having a serious or unstable medical condition, including cardiovascular, hepatic, endocrinologic, neurological or renal conditions.
* Clinically significant abnormalities on laboratory or ECG exams or those which, in the investigator ́s opinion, indicate a serious medical issue, require a major intervention or may interfere in the antidepressant treatment, also constitute grounds for exclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Early Improvement | 2 Weeks
  20% reduction of baseline score on the Hamilton Depression Scale (HAMD-17)

SECONDARY OUTCOMES:
Response | 4 and 8 weeks
  50% reductions of baseline score on the Hamilton Depression Scale (HAMD-17)
Remission | 8 and 24 weeks
  Score less than 7 points on the Hamilton Depression Scale (HAMD-17)

CONTACTS AND LOCATIONS:
Overall Officials: Moreno A Ricardo, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Insitute of Psychiatry of the University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Papakostas GI, Perlis RH, Scalia MJ, Petersen TJ, Fava M. A meta-analysis of early sustained response rates between antidepressants and placebo for the treatment of major depressive disorder. J Clin Psychopharmacol. 2006 Feb;26(1):56-60. doi: 10.1097/01.jcp.0000195042.62724.76. PMID 16415707
- [Background] Thase ME. Methodology to measure onset of action. J Clin Psychiatry. 2001;62 Suppl 15:18-21. PMID 11444762
- [Background] Szegedi A, Jansen WT, van Willigenburg AP, van der Meulen E, Stassen HH, Thase ME. Early improvement in the first 2 weeks as a predictor of treatment outcome in patients with major depressive disorder: a meta-analysis including 6562 patients. J Clin Psychiatry. 2009 Mar;70(3):344-53. doi: 10.4088/jcp.07m03780. Epub 2009 Feb 24. PMID 19254516
- [Derived] Carneiro AM, Pereira DA, Fernandes F, Baptista MN, Brunoni AR, Moreno RA. Distorted thoughts as a mediator of depressive symptoms in patients with major depressive disorder: a longitudinal study. Health Qual Life Outcomes. 2023 Aug 14;21(1):88. doi: 10.1186/s12955-023-02178-y. PMID 37580739